CLINICAL TRIAL: NCT07282236
Title: Quality of Reduction, Position of the Lag Screw and Mechanical Complications in Unstable Interthrochanteric Hip Fractures. A Comparison Between Gamma and InterTAN Nail.
Brief Title: Retrospective Comparative Outcomes of Gamma and InterTAN Nail for Unstable Intertrochanteric Hip Fractures
Status: Completed | Type: Observational
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Other Study IDs: UCV/2022-2023/009
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Unstable Throchanteric Hip Fractures; Pertrochanteric Fracture of Femur
Keywords: Throchanteric Fractures; Gamma nail; InterTAN nail
MeSH Terms: interventions — Fracture Fixation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Gamma Nail Group: The Gamma Nail Group consists of patients diagnosed with unstable trochanteric fractures who underwent surgical management using a Gamma cephalomedullary nail. This intervention involves internal fixation with a short or long intramedullary device designed to provide stable biomechanical support for unstable peritrochanteric fracture patterns. Patients in this group received the Gamma nail as the primary method of fracture stabilization, with the goal of achieving early mobilization, maintaining fracture alignment, and reducing the risk of mechanical complication.
  Interventions: Device: Fracture fixation with cephalomedullary nails
- InterTAN Nail Group: The InterTAN Nail Group includes patients with unstable trochanteric fractures who were treated surgically using an InterTAN cephalomedullary nail. This intervention consists of internal fixation with a dual integrated screw intramedullary device designed to enhance rotational and axial stability in unstable peritrochanteric fracture patterns. Patients in this group received the InterTAN nail as the primary method of fracture stabilization, aiming to improve construct rigidity, facilitate early mobilization, and support optimal fracture healing.
  Interventions: Device: Fracture fixation with cephalomedullary nails

INTERVENTIONS:
Device: Fracture fixation with cephalomedullary nails — No differences with the routine surgery for trochanteric fractures

SUMMARY:
Objective: compare outcomes of unstable intertrochanteric hip fractures treated with two commercially available implants. Design: retrospective observational cohort of 288 treated with a Gamma® nail and 398 with an InterTAN® nail. Patients were operated between 1997 and 2010. Primary outcomes: satisfactory reduction, optimal cephalic screw placement, and to evaluate the incidence of mechanical complications; secondary measures included the tip-apex distance (TAD), hematocrit (Hto) and hemoglobin (Hb) drop, transfusion requirement and volume, hospital length of stay and the time to first ambulation.

DETAILED DESCRIPTION:
Rationale: to evaluate whether outcomes differ between two commonly used cephalomedullary nails for unstable intertrochanteric hip fractures in routine practice.

Setting: double-centre, single-city retrospective cohort with consecutive patients treated by the same surgeon-Gamma2® at the Hospital Clínico Universitario (1997-2002; n=288) and InterTAN® at Vithas Hospitals (2002-2010; n=398). Cohorts: defined by the implant used in usual care; adults ≥65 years with unstable AO/OTA A2-A3 patterns were included; key exclusions were stable patterns, pathologic fractures, subtrochanteric extension, poor radiographs, and <6-month follow-up. Planned analyses: between-group comparisons of reoperation and implant-related complications (primary focus), plus perioperative and functional parameters, using χ²/t-tests as appropriate adjusting for age, sex, ASA class, AO/OTA pattern, reduction quality, and screw position metrics (e.g., TAD); results reported as effect sizes with 95% CIs, with sensitivity analyses by fracture pattern and reduction quality

ELIGIBILITY:
Inclusion Criteria:

* Unstable trochanteric fractures confirmed radiographically according to OTA (Orthopedic Trauma Association), treated with Gamma or InterTAN nail,
* available follow-up for ≥ 6 months

Exclusion Criteria:

* Pathological fractures
* Polytrauma precluding standard treatment/follow-up
* Missing key variables/outcomes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who received the Gamma nail (288) underwent surgery at the Hospital Clínico Universitario, Valencia (1997-2002). On the other hand, the patients operated upon the InterTAN nail (398) underwent surgery at the Vithas Hospitals Group in Valencia between January 2002 and December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Implant-related complications | 6 months
  Incidence of device-related adverse events (e.g., cut-out, varus collapse).

SECONDARY OUTCOMES:
Quality of fracture reduction | Immediately postoperative (within 24 hours)
  Satisfactory or unsatisfactory according to Baumgaertner's criteria
Cephalic screw placement | Immediately postoperative (within 24 hours)
  Position of the lag screw according to Cleveland-Bosworth quadrants

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine and Health Sciences, Valencia Catholic University, Valencia, VALÈNCIA, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Núñez JH, Moreira F, Surroca M, Martínez-Peña J, Jiménez-Jiménez MJ, Ocrospoma-Flores B, Castillón P, Guerra-Farfán E. Hip fractures in Spain. How are we? Systematic review and meta-analysis of the published registries. Rev Esp Cir Ortop Traumatol. 2024 Oct 16:S1888-4415(24)00156-5. English, Spanish. doi: 10.1016/j.recot.2024.09.010. Epub ahead of print. PMID: 39419269.
- [Result] Werner M, Macke C, Gogol M, Krettek C, Liodakis E. Differences in hip fracture care in Europe: a systematic review of recent annual reports of hip fracture registries. Eur J Trauma Emerg Surg. 2022 Jun;48(3):1625-1638. doi: 10.1007/s00068-021-01797-8. Epub 2021 Oct 8. PMID 34623474
- [Result] Shankar KN, Li A. Older Adult Falls in Emergency Medicine, 2023 Update. Clin Geriatr Med. 2023 Nov;39(4):503-518. doi: 10.1016/j.cger.2023.05.010. Epub 2023 Jul 6. PMID 37798062
- [Result] Kalan Farmanfarma K, Yarmohammadi S, Fakharian E, Gobbens RJ, Mahdian M, Batooli Z, Lotfi MS, Abedzadeh-Kalahroudi M, Vatan RF, Khosravi GR, Fazel MR, Sehat M. Prognostic Factors of Hip Fracture in Elderly: A Systematic Review. Int J Prev Med. 2024 Aug 30;15:42. doi: 10.4103/ijpvm.ijpvm_169_23. eCollection 2024. PMID 39381356